CLINICAL TRIAL: NCT04015661
Title: Induction Chemotherapy With Nab-paclitaxel and Nedaplatin Followed by Concurrent Chemoradiotherapy in Patients With Locally Advanced Nasopharyngeal Carcinoma
Brief Title: Induction Chemotherapy Followed by Concurrent Chemoradiotherapy in Patients With LA-NPC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fuzhou General Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20190515
Record Dates: First submitted 2019-07-09; First posted 2019-07-11 (Actual); Last update posted 2019-07-11 (Actual); Status verified 2019-07

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — 130-nm albumin-bound paclitaxel; Paclitaxel; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nab-paclitaxel+Nedaplatin (Experimental): induction chemotherapy by nab-paclitaxel and nedaplatin followed by concurrent chemoradiotherapy
  Interventions: Drug: Nab-paclitaxel
- Paclitaxel+Nedaplatin (Active Comparator): induction chemotherapy by paclitaxel and nedaplatin followed by concurrent chemoradiotherapy
  Interventions: Drug: Nab-paclitaxel

INTERVENTIONS:
Drug: Nab-paclitaxel — induction chemotherapy with nab-paclitaxel and nedaplatin followed by concurrent chemoradiotherapy
  Other Names: Paclitaxel for Injection (Albumin Bound)

SUMMARY:
Nasopharyngeal carcinoma (NPC) is a malignant tumor that originates in nasopharyngeal epithelial cells. It is common in southern China and Southeast Asia, but the incidence rate is low in most parts of the world. According to the World Health Organization survey, 80% of nasopharyngeal carcinomas occur in China, with high incidence in southern China, as high as 30-50/100,000, such as Guangdong, Guangxi, Hunan, and Fujian. In 2015, Chinese cancer statistics showed that there were about 60,600 new cases of nasopharyngeal carcinoma in China, and the number of deaths was about 34,100. Radiation therapy is the main treatment for nasopharyngeal carcinoma. Early stage I and IIa achieved a 5-year survival rate (OS) of 90% and 84%, respectively . However, the treatment outcomes of most patients with locally advanced nasopharyngeal carcinoma are not ideal.

ELIGIBILITY:
Inclusion Criteria:

1. Age, 18-75 years old.
2. Patients with newly histologically confirmed NPC.
3. WHO Type Ⅱ and Ⅲ.
4. Tumor staged as Ⅲ-ⅣA (according to the 8th AJCC edition).
5. No serious organ dysfunction of heart, lung, liver, kidney.
6. No distant metastasis.
7. Hematological examinations:WBC≥3.5×109/L, NEUT#≥1.5×109/L, PLT≥90×109/L, HB≥90g/L.
8. Normal liver function test：Alanine Aminotransferase (ALT)、Aspartate Aminotransferase (AST) <1.5×upper limit of normal (ULN) concomitant with alkaline phosphatase (ALP) ≤2.5×ULN, and bilirubin ≤1.5×ULN，creatinine clearance ≥60 ml/min.
9. Patients must be given written informed consent.

Exclusion Criteria:

1. age >75 years or <18years.
2. Prior chemotherapy or surgery (except diagnostic) to primary tumor or nodes.
3. History of previous radiotherapy and chemotherapy.
4. Known or suspected to be allergic to platinum and Nab-paclitaxel.
5. Pregnancy or lactation.
6. Any severe intercurrent disease, which may bring unacceptable risk or affect the compliance of the trial.
7. Peripheral sensory neuropathy> grade 1.
8. Uncontrolled heart clinical symptoms or diseases.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2019-07-09 (Estimated); Primary Completion 2020-12-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 3 years
  To be determined by measurement of target lesions according to RECIST criteria

SECONDARY OUTCOMES:
Progression-Free Survival(PFS) | 3 years
  From the date of enrollment to the date of either locally, regionally or distant failure or last follow-up
Overall survival（OS） | 3 years
  From the date of enrollment to the date of death is observed or to last follow-up visit

CONTACTS AND LOCATIONS:
Overall Officials: zhichao fu, M.D, Study Chair — Fuzhou General Hospital of Nanjing Military Regio，Department of Radiotherapy
Locations (1):
- No. 156, North Road, Xierhuan Road, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No